CLINICAL TRIAL: NCT05869942
Title: Histological and Histochemical Study of Vitiligo Pathogenesis in Sohag University Hospital Patients
Brief Title: Histochemical Study of Vitiligo in Sohag University Hospital Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Mamdouh Ahmed, Demonstrator at Histology and cell Biology department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-04-25MS
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Vitiligo
Keywords: vitiligo; autoimmunity; apoptosis; melanocytes
MeSH Terms: conditions — Vitiligo; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Under complete sterile precautions, Skin biopsy will be taken from healthy volunteers of the control group via 3 mm disposable punches and two biopsies will be taken from patients with vitiligo, one from vitiligenous lesion and another from normal skin then will be rinsed in physiological saline and fixed in formalin for 24 hours. The preserved tissues will be trimmed for processing, then undergo dehydration with ethyl alcohol, clearing with xylene, infiltration and embedding with paraffin wax. Paraffin wax blocks will be sectioned at 5μ then mounted on glass slides. Sectioned slides will be stained with hematoxylin and eosin and other histological stains and mounted with (DPX). And examined by light microscope.
  The pathological changes in vitiligenous skin will be detected. Monoclonal HMGB1 and active caspase 3 antibodies assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- groupA (Diseased group) (Active Comparator): patients with Vitiligo
  Interventions: Diagnostic Test: Light microscopic studies; Diagnostic Test: Immunohistochemical studies
- group B(Control group) (Active Comparator): Normal control group not diseased
  Interventions: Diagnostic Test: Light microscopic studies; Diagnostic Test: Immunohistochemical studies

INTERVENTIONS:
Diagnostic Test: Light microscopic studies — Under complete sterile precautions, Skin biopsy will be taken from healthy volunteers of the control group via 3 mm disposable punches and two biopsies will be taken from patients with vitiligo, one from vitiligenous lesion and another from normal skin then will be rinsed in physiological saline and fixed in formalin for 24 hours. The preserved tissues will be trimmed for processing, then undergo dehydration with ethyl alcohol, clearing with xylene, infiltration and embedding with paraffin wax. Paraffin wax blocks will be sectioned at 5μ then mounted on glass slides. Sectioned slides will be stained with hematoxylin and eosin and other histological stains and mounted with (DPX). And examined by light microscope. The pathological changes in vitiligenous skin will be detected
Diagnostic Test: Immunohistochemical studies — Monoclonal HMGB1 and active caspase 3 antibodies

SUMMARY:
Vitiligo is a common acquired idiopathic disorder characterized by depigmentation of the skin, hair, and mucous membranes in the form of macules and patches due to selective melanocyte destruction . Incidence of Vitiligo is about 0.5% to 2% of the world's population, and its incidence continues to increase. Vitiligo can appear at any age group especially in the second and third decades of life. About one-third of vitiligo patients are children under ten years old Vitiligo can be classified into non-segmental, segmental, mixed and unclassifiable/undetermined types. Vitiligo has a negative impact on patient's quality of life by decreasing their self-confidence and causing significant psychological distress.

DETAILED DESCRIPTION:
The pathogenesis of vitiligo is still unclear but some theories can explain it such as oxidative stress, autoimmunity, autocytotoxicity, genetic factors, neural and melanocytorrhagy . Loss of pigment which occur in vitiligo may be due to two main causes: absence of melanocytes and/or the inability of melanocytes to produce and store melanin in melanosomes in the process of melanogenesis.

High mobility group box protein B1 (HMGB1) normally presents in the nucleus to maintain genomic stabilization and regulate gene transcription. but, HMGB1 can be released outside the cell due to exposure to stressful factors such as oxidative stress and function as a damage-associated molecular pattern (DAMP) protein leading to strong proinflammatory effects. Recent data showed that HMGB1 is overexpressed in both blood and lesional specimens from vitiligo patients. Moreover, oxidative stress triggers the release of HMGB1 from keratinocytes and melanocytes, indicating that HMGB1 may participate and play a crucial role in the pathological process of vitiligo.

HMGB1 Directly induces Melanocyte apoptosis through stimulation with reactive oxidative stress (ROS) or ultraviolet B (UVB) in vitro which significantly increases the release of HMGB1 from keratinocytes, which inhibits the expression of melanogenesis-related molecules such as microphthalmia- associated transcription factor (MITF), tyrosinase-related proteins and the gp100 protein in a paracrine manner and finally activate caspase-3 to trigger melanocyte apoptosis

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with vitiligo aged 18-50 years old.

Exclusion Criteria:

* Pregnancy
* Lactation
* Patient on immunosuppressive treatment for vitiligo over the last month
* Skin diseases, other than vitiligo.
* Systemic diseases particulary endocrine disorders and autoimmune connective tissue diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of tissue expression of HMGB1 in patients with vitiligo compared to normal control. | 12 months
  Monoclonal HMGB1 antibodie assessment by Skin biopsy from healthy volunteers of the control group via 3 mm disposable punches and two biopsies will be taken from patients with vitiligo, one from vitiligenous lesion and another from normal skin.
Assessment of tissue expression of active caspase 3 in patients with vitiligo compared to normal | 12 months
  active caspase 3 antibodie assessment by Skin biopsy from healthy volunteers of the control group via 3 mm disposable punches and two biopsies will be taken from patients with vitiligo, one from vitiligenous lesion and another from normal skin.

CONTACTS AND LOCATIONS:
Overall Officials: Doha S Mohamed, professor, Study Chair — Sohag University, Faculty of Medicine; Zeinab A Goda, lecturer, Study Director — Sohag University, Faculty of Medicine
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellei B, Picardo M. Premature cell senescence in human skin: Dual face in chronic acquired pigmentary disorders. Ageing Res Rev. 2020 Jan;57:100981. doi: 10.1016/j.arr.2019.100981. Epub 2019 Nov 14. PMID 31733332
- [Background] Faraj S, Kemp EH, Gawkrodger DJ. Patho-immunological mechanisms of vitiligo: the role of the innate and adaptive immunities and environmental stress factors. Clin Exp Immunol. 2022 Jan 28;207(1):27-43. doi: 10.1093/cei/uxab002. PMID 35020865
- [Background] Wei G, Pan Y, Wang J, Xiong X, He Y, Xu J. Role of HMGB1 in Vitiligo: Current Perceptions and Future Perspectives. Clin Cosmet Investig Dermatol. 2022 Oct 13;15:2177-2186. doi: 10.2147/CCID.S381432. eCollection 2022. PMID 36267690
- [Background] Wang J, Pan Y, Wei G, Mao H, Liu R, He Y. Damage-associated molecular patterns in vitiligo: igniter fuse from oxidative stress to melanocyte loss. Redox Rep. 2022 Dec;27(1):193-199. doi: 10.1080/13510002.2022.2123864. PMID 36154894